CLINICAL TRIAL: NCT00561275
Title: Phase 1 Study of Multiple Peptide Vaccine Therapy and GM-CSF in Treating Patients With Esophageal Cancer
Brief Title: Safety Study of Multiple Peptide Vaccine to Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Japanese Foundation for Cancer Research (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB-454
Record Dates: First submitted 2007-11-14; First posted 2007-11-20 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — LY6K protein, human; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: LY6K, VEGFR1, VEGFR2 — 1 mg/body every two week with GM-CSF, 4 cycles

SUMMARY:
This is a phase 1 study of multiple peptide vaccine therapy and GM-CSF in treating patients with esophageal cancer.

DETAILED DESCRIPTION:
LY6K (lymphocyte antigen 6 complex, locus K) was identified as a new target of tumor associated antigen using cDNA microarray technologies combined with the expression profiles of normal and cancer tissues. On the other hand, anti-angiogenic therapy is now considered to be one of promising approaches to treat of cancer. In this clinical trial, we evaluate the safety and immune responses of multiple peptide cocktail including LY6K and vascular endothelial growth factor receptor 1 (VEGFR1) and vascular endothelial growth factor receptor 2 (VEGFR2) together with IFA and GM-CSF as immunoadjuvants in patients who had LY6K expressed primary esophageal cancer. Toxicity profiles will be monitored, and antigen specific T cell responses will be described.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have metastatic disease of esophageal cancer, and treatment has failed, or in the situation where effective therapy is not available, or has been refused due to severe adverse effects of chemotherapy
2. WHO performance status of 0 to 2
3. Age ≥ 20 years, ≤75 years
4. Chemotherapy, any type of radiation therapy, or immunotherapy within 4 weeks before study entry
5. Expected survival of at least 3 months
6. WBC≥ 2,000/mm³ Platelet count ≥ 100,000/mm³ Total bilirubin ≤ 1.5 x the institutional normal upper limits AST, ALT, ALP ≤ 2.5 x the institutional normal upper limits Creatinine ≤ 1.5 x the institutional normal upper limits
7. Patients must be HLA-A2402
8. Primary lesion of esophageal cancer must express LY6K
9. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Serious infections requiring antibiotics
4. Patient with peptic ulcer disease
5. Previous history of intestinal perforation
6. bleeding disorders (INR ≥ 1.5)
7. Necessity of drug-mediated inhibition with platelet function
8. Taking antithrombogenic agents within 10 days
9. Serious hypertension
10. Previous history of arterial thrombosis or venous thrombosis
11. Other malignancy within 5 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ
12. Clinically significant heart disease or previous history of myocardial infarction within the past 12 months
13. Concomitant treatment with steroids or immunosuppressing agent
14. Disease to the central nervous system
15. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Toxicity of multiple peptide vaccinations | one year

SECONDARY OUTCOMES:
Immune responses including LY6K, VEGFR1 and VEGFR2 specific T cells | one year

CONTACTS AND LOCATIONS:
Overall Officials: Takuya Takayama, M.D.Ph.D, Principal Investigator — Cancer Institute of Japanese Foundation for Cancer Research
Locations (1):
- Takuya Takayama M.D.Ph.D, Tokyo, Japan

REFERENCES:
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873